CLINICAL TRIAL: NCT00314431
Title: Randomized Comparison of Two Models of Post-NICU Care for Preterm Infants With Neonatal Chronic Lung Disease
Brief Title: Post-hospitalization Nursing Effectiveness (PHONE) Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BG99547; R01HS007928 (AHRQ)
Record Dates: First submitted 2006-04-11; First posted 2006-04-13 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2006-04

CONDITIONS: Bronchopulmonary Dysplasia; Prematurity
Keywords: neonatal chronic lung disease; bronchopulmonary dysplasia; prematurity; telephone follow up; care coordination; children with special health care needs
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth

INTERVENTIONS:
Procedure: Care coordination by telephone contacts with a nurse

SUMMARY:
Based on success with telephone follow up for other groups of medically fragile infants, we designed an innovative model of post-hospital comprehensive and coordinated follow-up for infants with chronic lung disease. In this model, which we refer to as community-based follow-up, medical management was coordinated by a nurse specialist, through frequent telephone contacts with the infants' primary caregiver. This model of follow up care was compared, in a randomized trial, with the more traditional model - multidisciplinary medical center-based care. We hypothesized that community-based care would lead to health and developmental outcomes similar to those observed with center-based care.

DETAILED DESCRIPTION:
METHODS Study design A randomized equivalence trial was designed to compare community-based follow up with medical-center based follow up. The primary outcome was assessed at one year adjusted age.

Study participants Infants were recruited in five neonatal intensive care units in northwest North CArolina. These were the only sites providing neonatal intensive care in a twenty-county region in northwest North Carolina. Infants were born between March 1996 and September 1999. Infants were eligible for the study if they were born before 33 weeks gestational age, required supplemental oxygen at 36 weeks gestational age, and were discharged home after neonatal intensive care. Neonates who had major congenital anomalies and/ or had tracheostomy tubes were excluded. Also excluded were families in which the mother did not speak English, because the intervention depended on verbal communication with the nurse specialist, and families who lived more than 150 miles from our clinic because such families typically are referred to regional neonatal center closer to their home.

Randomization A randomization list was prepared by a biostatistician who was not involved in data collection or clinical care of the infants. Lists of randomization assignments, which were kept in a sealed envelope in a locked drawer, were prepared for each of the five sites at which participants were recruited. Randomization assignments were made in blocks sizes of two and four. Once a study participant arrived home from the neonatal intensive care unit, a research assistant uncovered the next assignment on the randomization list, which was kept in a sealed envelope in a locked drawer.

Intervention If the family did not have telephone service at the time of the infant's discharge, a telephone was installed at no cost to the family, within one week of the infant's discharge from the hospital. Research funds were used to reimburse all families for the cost of local phone service for the duration of the study. Families assigned to either intervention could contact the nurse specialist on a toll-free long distance line with voice mail which recorded messages when the phone was not attended.

The intervention team consisted of two neonatologists, a pediatric social worker, and a nurse specialist.

Community-based follow up Telephone contacts were made to the infants' primary caregiver by the nurse specialist twice weekly in the first month after discharge, weekly in months two through four, and monthly thereafter until the infant attained 12 months adjusted age. At each telephone contact, the nurse used a semi-structured format to inquire about the infant's health, community resources utilized by the infant, and potential stressors and sources of support for the family. She also inquired about the infant's medications and feedings. If she judged the infant would benefit from a change in medical management, additional assessments or a subspecialty referral, she discussed the proposed change with one of the two study neonatologists. If there was agreement, the recommendation was communicated to the family and the infant's primary care provider. The nurse specialist also coordinated care for the infant by communicating with home health nurses, public health nurses, early intervention specialists, physical therapists, and pediatric sub-specialists.

Medical center-based follow up For infants who were discharged home on supplemental oxygen, the nurse specialist made a home visit 1 to 2 weeks after discharge. During this visit, the nurse specialist obtained interim medical history, performed physical assessment including pulse oximetry and body weight, reviewed discharge instructions regarding medication dosage and use of durable medical equipment, and answered caregiver's questions about the infant's care. If the nurse specialist had concerns about the medical condition of the infant, she made changes to the plan of care after consultation with the study neonatologist.

All infants assigned to the center-based care group were seen in the regional, high-risk infant multidisciplinary clinic at Wake Forest University School of Medicine. The first clinic visit occurred approximately one month after their discharge. A multidisciplinary team consisting of the social worker, the nurse specialist and the neonatologist obtained detailed interim medical history (feeding, respiratory status, medication history, illnesses and health-services utilization) and performed a complete physical examination. Family stressors and resources were discussed. All infants were scheduled for visits at four, eight, and twelve months adjusted age. In addition, infants who were using supplemental oxygen were seen at an interval of 1-2 months until all of the following criteria were met: 1) their growth rate was 15-30 grams/day, 2) they were no longer using supplemental oxygen or other medications, and 3) they were no longer using a home apnea monitor. At each clinic visit, the infant and parent or guardian were seen individually by the clinic social worker, the nurse specialist for this project, and one of the two neonatologists who conferred as a group and developed a plan of care. This plan was communicated to the family by the nurse specialist.

Communication with primary care providers Within 24 hours after randomization, the principal investigator called the infants' primary care providers to inform them about the study design and that the parents have consented to participate in the study. In the case of infants randomized to community-based care, the primary care provider was given the choice of making the decisions about changes in medical care independently or jointly with the nurse specialist. A copy of a protocol for management of infants with CLD, developed by the study team was mailed to each primary care provider. After each clinic visit (for the center-based group) the primary care provider received a letter describing findings, impressions, and recommendations. Contacts with the primary care physicians of infants randomized to community-based care occurred whenever the nurse specialist believed that a change in care was indicated.

Outcomes assessed during the first year Self-administered questionnaires were used to assess psychosocial status of the family, healthcare utilization and healthcare expenses at baseline, one, four, seven and eleven months. Each time the family completed study questionnaires and when home visits were made, families were given twenty dollars as compensation. At eleven months, a research assistant conducted a home visit and assessed the home using the Caldwell HOME Inventory,27 and the parent-infant interaction using a scale developed by Holditch and Miles.28 Only results of rehospitalization rates during the first year will be presented in this paper.

Outcomes assessed at one year adjusted age All children were evaluated at one year adjusted age at a Development Evaluation Clinic dedicated solely to developmental assessments of high-risk infants. The primary outcome, the Bayley Scales of Infant Development-Second Edition (BSID-2) Mental Developmental Index (MDI)I, and two secondary outcomes - the BSID Pyschomotor Developmental Index (PDI) and the Vineland Adaptive Behavioral Scales (VABS) were assessed by child psychologists or psychology graduate students supervised by a child psychologist, who were not aware of the child's intervention group or medical history. After the testing was completed, the psychologist was informed of the infant's gestational age at birth, so that the BSID scores could be corrected for the degree of prematurity. The BSID MDI is a widely used and validated developmental assessment tool to measure cognitive development in the first two years of life. The BSID PDI measures fine and gross motor development.29 The population mean for both the scores is 100 with a standard deviation of 15. Higher score on BSID MDI and PDI represents better cognitive and motor functioning respectively.30 When the BSID MDI/ PDI score was less than 50, then the score was extrapolated as described previously.31

The Vineland Adaptive Behavior Scales are a parent-reported measure of child adaptive development. The scale assesses four domains of adaptive development: communication, daily living skills, socialization, and motor skills. The overall Adaptive Behavior Composite (ABC) is a standard score based on the child's age, with higher scores representing better adaptive functioning. Population mean for ABC is 100 and the standard deviation is 15.32

Anthropometric measurements were performed by a neonatologist, who was aware of the infants' intervention assignment, using a pediatric scale for weight, a length board for length, and a tape measure for head circumference. Growth delay was defined as weight for length less than 5th percentile at one year adjusted age. At 1 year follow-up, a research assistant reviewed each child's clinic chart and noted whether any of the following health conditions or receipt of health-services: cerebral palsy, blindness, hearing impairment, seizure disorder, oxygen requirement, need for tracheostomy tube and ventriculo-peritoneal shunt.

ELIGIBILITY:
Inclusion Criteria:

* Infants were eligible if they were born before 33 weeks gestational age, required supplemental oxygen at 36 weeks gestational age, and were discharged home after neonatal intensive care.

Exclusion Criteria:

* Neonates who had major congenital anomalies and/ or had tracheostomy tubes were excluded. Also excluded were families in which the mother did not speak English, because the intervention depended on verbal communication with the nurse specialist, and families who lived more than 150 miles from our clinic because such families typically are referred to regional neonatal center closer to their home.

Ages: 1 Day to 483 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150
Dates: Start 1996-05; Study Completion 2000-08

PRIMARY OUTCOMES:
Bayley Scales of Infant Development-Second Edition

SECONDARY OUTCOMES:
Growth through one year of age
Rehospitalizations in the first year of life
Vineland Adaptive Behavioral Scales

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M O'Shea, MD, MPH, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University School of Medicine, Winston-Salem, North Carolina, United States